CLINICAL TRIAL: NCT02529163
Title: Evaluating the Efficacy of a Late-Life Schizophrenia Integrated Care Pathway to Treat Acute Psychotic Symptoms
Acronym: LLS-ICP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Petal Abdool, Staff Psychiatrist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 032/2015
Record Dates: First submitted 2015-08-11; First posted 2015-08-20 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Integrated Care Pathway; Acute Psychotic Episode; Randomised Control Trial
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Late-life Schizophrenia ICP (Active Comparator): The Late-Life Schizophrenia ICP arm will follow a medication algorithm composed of 3 trials and titration schedule with prompts.
  First trial is Risperidone (2- 4mg daily).
  Second trial: Quetiapine (100 - 400mg daily) OR Aripiprazole (100 - 200mg daily) OR OR Ziprasidone (80mg daily) OR Loxapine (100mg daily)
  Third trial: Clozapine (450mg daily) or Olanzapine (20mg daily)
  If non compliant depot preparation of: Paliperidone (50 - 150mg monthly), Risperidone (12.5 - 50mg q 2 weeks), Flupentixol (10 - 20mg q 2-3 weeks) or Aripiprazole ( up to 400mg monthly)
  Prompts will be given to for non-pharmacological interventions such as:
  * metabolic monitoring
  * skin hygiene
  * pain management
  * nutritional counseling
  * counseling
  Interventions: Other: Late-life Schizophrenia ICP
- Treatment as Usual (TAU) (Active Comparator): The TAU will not receive any prompts to follow a specific treatment. The TAU group will be treated according to the current standard of care by the treating physician. They will have an opportunity to be offered the same non-pharmacological interventions seen with the ICP group but at the discretion of the treating physician. Pharmacological interventions will include an anti-psychotic medication that is selected at the discretion of treating physician with no set titration schedule or timeline to meet a maximum dosage. Max dosage will be decided by the treating physician.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Late-life Schizophrenia ICP — The ICP medication algorithms first trial begins with:
  * Risperidone titrated to a max dose
  Failure to Risperidone will lead to a second trial with either:
  * Quetiapine OR Aripiprazole
  If subject refuses or if this trial does not work, then offer:
  * Ziprasidone or Loxapine
  Failure of 2 anti-psychotic trials results in:
  * Clozapine trial
  If subject refuses a Clozapine trial then:
  * Olanzapine offered
  titrations occur over 33-36 day period (inpatient) or 12 week period (out patient) with each 0.5 mg titration after the target dose requiring a CGI-E
  If compliance is an issue then a depot preparation:
  * Paliperidone
  * Risperidone
  * Flupentixol
  * Aripiprazole
  Physicians will be prompted for non-pharmacological interventions
  Other Names: LLS-ICP; Late-life Schizophrenia Integrative Care Pathway
  Arms: Late-life Schizophrenia ICP
Other: Treatment as Usual — The TAU group will be offered non-pharmacological interventions such as (but not limited to):
  * metabolic monitoring
  * skin hygiene
  * pain management
  * nutritional counseling
  * family counselling
  * Financial/housing support
  * Group CBT (Cognitive Behavioral Therapy)
  Physicians treating this group will use their own discretion as they will not be prompted like the ICP group.
  Pharmacological interventions contain anti-psychotic medication selected at the discretion of the treating physician provided it fall under the current standard of care such as:
  * Risperidone
  * Aripiprazole
  * Quetiapine
  * Olanzapine
  * Paliperidone
  * Clozapine
  * Ziprasidone
  Max dosing and the time to reach the target dose is done at the discretion of the treating physician.
  Other Names: TAU
  Arms: Treatment as Usual (TAU)

SUMMARY:
As of late Integrated Care Pathways (ICPs) have been shown to improve quality of care in the medical field with special attention given to mental health in particular. One aspect of metal health that has not seen the incorporation of ICPs is in the area of schizophrenia. Late life Schizophrenia (LLS) is defined as suffering from schizophrenia and being 50 years of age or older. The LLS-ICP study will look at the efficacy of an ICP in late life schizophrenia versus treatment as usual (TAU). Participants with LLS and having psychotic symptoms above a predefined threshold will be randomly assigned to a TAU group or an ICP group. The primary outcome measure will be reduction in symptom severity as measured by clinical global impression severity scale (CGI-S) and brief psychiatric rating scale (BPRS). If successful, this study will provide strong evidence to implement LLS-ICP across different inpatient and outpatient settings.

DETAILED DESCRIPTION:
This study aims to investigate whether a Late-Life Schizophrenia-Integrated Care Pathway (LLS-ICP) is superior to treatment as usual (TAU) in the treatment of psychotic symptoms of patients with schizophrenia or schizoaffective disorder. The investigators hypothesize that the LLS-ICP will be superior to TAU and result in 1.higher rates of response, 2. shorter times to response, 3. less side effects, 4. and better functional outcomes. The LLS-ICP study will be the first randomized controlled study to assess the efficacy of an ICP in patients with schizophrenia or schizoaffective disorder in this region. If successful, it will lead to the development of new and innovative approaches to health care delivery to patients with chronic schizophrenia or schizoaffective disorder not just within this institution but also at other sites in the community. The nature of ICPs as algorithmic and systematic in providing assessments and treatments render them ideal to be disseminated to medical practice outside of the institution of where they have been developed. These settings can include primary care clinics, supportive living environments, and long-term care homes where patients with chronic schizophrenia or schizoaffective disorder are being cared for.

ELIGIBILITY:
Inclusion Criteria:

* All races and ethnicity
* Meets DSM-IV TR (Diagnostic and Statistical Manual Version 4 Text Revision) criteria for a current diagnosis of Schizophrenia
* clinically unstable and in an acute episode as defined by a CGI severity score greater than 3 or a BPRS thought disorder sub-scale score higher than 6 (total score).
* Willingness and ability to speak English
* Willingness to provide informed consent or has a proxy who can do so
* Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria:

* Diagnosis of bipolar disorder, current major depressive episode or an acutely psychotic episode secondary to a non-schizophrenic disorder
* Meets diagnostic criteria for substance use or dependence within the 6 months prior to the initial assessment except for caffeine or nicotine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of LLS-ICP using a medication algorithm and evaluating with the clinical global impression severity scale (CGI-S) and brief psychiatric rating scale (BPRS) | 18 months
  Reduction in symptom severity will be measured using CGI-S (1 item 7 point scale with 0 being not assessed and 7 being most extremely ill patient) and (BPRS) which will be used to measure psychiatric symptoms such as hallucinations, anxiety or depression. ( 24 question scale rated from 0 being not assessed and 7 being extremely severe). Both scores will be aggregated to determine the reduction in overall symptoms and their severity in relationship to ICP and TAU groups.

SECONDARY OUTCOMES:
Efficacy of an Integrated Care Pathway on rate and time of response needed to treat acute psychotic episode measured by CGI-E for therapeutic response and global improvement. | 18 months
  Reduction in the rate and time to respond to medication during an acute psychotic episode measured by Clinical global impression - efficacy scale (4 item scale rated from 0 - 4 points with 0 being not assessed and 4 representing side effects outweighing therapeutic effect). This scale will be used to measure the efficacy of therapeutic response to the medication algorithm in the ICP against the standard treatment of care (TAU).
Efficacy of an Integrated Care Pathway on side effect burden using Simpson Angus Scale (SAS), Barnes Akathisia Scale (BAS/BARS), and Abnormal Involuntary Movement Scale (AIMS). | 18 months
  Reduction in the number and severity of medication side effects on participants. The SAS is a 10 item scale (0 stands for normal - 4 stands for exaggerated symptoms) used to assess Parkinsonian and extra-pyramidal side effects. BAS is a 4 item scale used to assess the severity of drug induced akathisia. AIMS is a 12 item scale (0 for normal - 4 for severe) used to assess dyskinesias. These scores will be aggregated to measure the side effect burden seen with use of atypical anti-psychotic medication used to treat schizophrenia. These scores will compare the side effect burden of the TAU group against the ICP group.
Efficacy of an Integrated Care Pathway on functional outcome using the Multnomah Community Ability Scale (MCAS) for social functioning and Montreal Cognitive Assessment scale (MoCA) to test for cognition. | 18 months
  Increase in functional outcome to be assessed using the MCAS which measures adaptive functioning including health, adjustment to living, social competence and behavioral problems. It is a 17 item scale which graded from 1-6 where 1 represents extreme impairment, 5 represents normal and 6 representing unknown. The MoCA is a cognitive test that contains 12 items and is scored on a 30 point scale where 30 represents excellent cognitive function and 0 represents very poor cognitive function. Both scales will be aggregated to determine the relationship of the ICP and TAU to functional outcomes by measuring both cognitive and social functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Petal Abdool, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We do plan to share individual data at the completion of the study. Data will be shared only if the participant has agreed to do so as indicated on their informed consent document. Data that is expected to be shared will include all assessments from each visit, time to relapse, and which arm of the study each participant is affiliated with. In addition, research data gathered as part of this study may be shared and provided to investigators affiliated with GMHS (or other secondary investigators ) for the purpose of conducting secondary analyses about late-life mental illness. If subjects are enrolled in multiple studies in GMHS, their research data will be shared across studies to reduce participant burden and avoid duplication of procedures.

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research